CLINICAL TRIAL: NCT00600964
Title: A Multi-Center, Open-Label, Phase I/II Study of Single-Agent GX15-070MS Administered Every 2 to 3 Weeks to Patients With Previously-Treated Chronic Lymphocytic Leukemia (CLL)
Brief Title: A Phase I/II Study of GX15-070MS in Untreated CLL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gemin X (Industry)
Responsible Party: Jean Viallet, MD, Gemin X, Inc.
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GX004
Record Dates: First submitted 2008-01-15; First posted 2008-01-25 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; obatoclax
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — obatoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GX15-070MS (Experimental): GX15-070MS at various doses and schedules
  Interventions: Drug: GX15-070MS

INTERVENTIONS:
Drug: GX15-070MS — A 60-minute or 3-hour IV infusion every 2-3 weeks.
  Other Names: Obatoclax
Drug: GX15-070MS — GX15-070MS at various doses and schedules
  Other Names: Obatoclax

SUMMARY:
This protocol is being run to determine the best phase II dose and schedule of obatoclax in patients with previously untreated CLL.

DETAILED DESCRIPTION:
Both 1 hour and 3 hour infusions of obatoclax every 3 weeks will be evaluated in ascending doses.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed B-CLL
* Previous standard systemic chemotherapy, including fludarabine. There are no limitations on additional, allowable type and amount of prior therapy. Acute toxicities from prior therapy must have resolved to ≤Grade 1
* Age ≥18 years
* ECOG Performance Status ≤1
* Life expectancy of >8 weeks

Exclusion Criteria:

* Patients receiving any other investigational agents (e.g., under another IND) or commercial agents or therapies administered with the intent to treat their malignancy
* Patients with history of seizure disorders
* Pregnant women and women who are breast feeding
* HIV-positive patients receiving combination anti-retroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-09; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Determine the recommended Phase II dose of GX15-070MS administered as a 60-minute and/or 3-hour infusion every 2 to 3 weeks | 14 days

SECONDARY OUTCOMES:
Estimate the response rate of previously-treated patients with CLL at the recommended Phase II dose of GX15-070MS administered as a 60-minute and/or 3-hour infusion every 2 to 3 weeks. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean Viallet, MD, Study Director — Gemin X, Inc.
Locations (5):
- United States (4):
  - University of CA- San Diego, La Jolla, California
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Milton S Hershey Medical Center Penn State Cancer Institute, Hershey, Pennsylvania
  - UT MD Anderson Cancer Center, Houston, Texas
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] O'Brien SM, Claxton DF, Crump M, Faderl S, Kipps T, Keating MJ, Viallet J, Cheson BD. Phase I study of obatoclax mesylate (GX15-070), a small molecule pan-Bcl-2 family antagonist, in patients with advanced chronic lymphocytic leukemia. Blood. 2009 Jan 8;113(2):299-305. doi: 10.1182/blood-2008-02-137943. Epub 2008 Oct 17. PMID 18931344